CLINICAL TRIAL: NCT01363830
Title: Short (2-weeks) Versus Long (6-weeks) Post-Operative Restrictions Following Lumbar Discectomy: A Prospective Randomized Control Study
Brief Title: Short Versus Long Post-Operative Restrictions Following Lumbar Discectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Bono, Christopher M. Bono, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009P001125
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Lumbar Disc Herniation
Keywords: Disc; lumbar; herniation
MeSH Terms: conditions — Intervertebral Disc Displacement; Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two-Week Post-Operative Restriction (Experimental): Restrict bending, lifting, and twisting for two-weeks following discectomy.
  Interventions: Behavioral: Two-Week Post-Operative Restriction
- Six-Week Post-Operative Restriction (Active Comparator): Restrict bending, lifting, and twisting for six-weeks following discectomy.
  Interventions: Behavioral: Six-Week Post-Operative Restriction

INTERVENTIONS:
Behavioral: Two-Week Post-Operative Restriction — Surgeon recommends the patient restrict bending, lifting, and twisting for two-weeks following discectomy.
  Arms: Two-Week Post-Operative Restriction
Behavioral: Six-Week Post-Operative Restriction — Surgeon recommends patient restrict bending, lifting, and twisting for six-weeks following discectomy.
  Arms: Six-Week Post-Operative Restriction

SUMMARY:
Post-operative restrictions following lumbar discectomy is a controversial topic. While the most widely accepted protocol restricts bending, lifting, and twisting for four to six weeks following discectomy, a number of studies support an early return to full activity without restriction. Since the goal of discectomy is to promptly provide pain relief and a return to a fully active lifestyle, perhaps post-operative restrictions are more hindering than beneficial.

Hypothesis: Post-operative restrictions following lumbar discectomy do not influence reherniation rate.

Specific Aim 1: To compare the reherniation rates between the 6-weeks of restriction and the 2-weeks of restriction groups.

Specific Aim 2: To determine the return to full activity and return to work dates of both the 6-weeks of restriction and 2-weeks of restriction groups.

Specific Aim 3: To assess the health outcomes of both the 6-weeks of restriction and 2-weeks of restriction groups.

DETAILED DESCRIPTION:
Upon enrollment, subjects will be randomized to the "6-weeks of restriction" or "2-weeks of restriction" group. Subjects will also be asked to provide/complete:

* demographical information
* VAS back and leg score
* Modified Oswestry questionnaire

All of the surgeries will be performed using a so-called limited discectomy in which the herniated disc fragment is removed without an aggressive disc space curettage. Prior to surgery, the subjects' discs will be classified by the Primary Investigator and Site Responsible Investigator on a T-2 weighted MRI according to the Carragee Disc Herniation Classification system.

The discs will be reassessed intraoperatively by the surgeon to confirm the assigned classification. In addition, a radiologist will review a random sampling set of discs on T-2 weighted MRI to eliminate bias and validate the classifications.

Subjects will be followed for a 2 year time period with study visits at 2 weeks, 6 weeks, 3 months, 1 year, and 2 years. At every follow-up visit, the following will be completed and/or documented:

* A reherniation (any clinical symptoms of a reherniation will be verified and documented by MRI)
* Return to full activity and/or work (date)
* VAS back and leg score
* Modified Oswestry questionnaire

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English speaking
* single level lumbar disc herniation
* surgical candidate
* no previous lumbar surgery
* primary radicular pain

Exclusion Criteria:

* Less than 18 years of age
* Non-English speaking
* Multi-level lumbar disc herniation
* Disc reherniation
* Previous lumbar surgery
* Primary low back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Reherniation Rates | 2 years
  To compare the reherniation rates between the restricted and unrestricted groups.

SECONDARY OUTCOMES:
Activity/Health Outcomes | 2 years
  To determine the return to full activity and return to work dates of both the restricted and unrestricted groups. Also, to assess the health outcomes of both the restricted and unrestricted groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Bono, M.D., Principal Investigator — Brigham & Women's Hospital / Harvard Medical School
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts